CLINICAL TRIAL: NCT06887062
Title: Dapagliflozin and Endothelin Receptor Antagonism in Large Vessel Vasculitis (DERAIL-LVV)
Acronym: DERAIL-LVV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC24184
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Large Vessel Vasculitis; Giant Cell Arteritis (GCA); Takayasu Arteritis
Keywords: Large vessel vasculitis; Takayasu arteritis; Giant cell arteritis; Endothelin; Bosentan; Inflammation; Endothelial dysfunction; Dual enodthelin receptor antagonism; dapagliflozin; SGLT2 inhibitor
MeSH Terms: conditions — Giant Cell Arteritis; Takayasu Arteritis; Inflammation | interventions — Bosentan; dapagliflozin

STUDY DESIGN:
Intervention Model Description: The study will incorporate both a prospective, case-control study and a nested prospective, open blinded study.
  Case-control study: this will be cross-sectional and assess endothelial function, arterial stiffness and 24-hour blood pressure in 30 patients with LVV in disease remission and 30 age-, sex- and cardiovascular risk factor-matched control subjects.
  Open-blinded study: This will be a 10-week open-blinded study in the same 30 subjects with LVV from the case-control study. All 30 participants will receive 6 weeks of bosentan and dapagliflozin, followed by 4 weeks of dapagliflozin. Outcomes will be measured at baseline, week 3, week 6 and week 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 participants with large vessel vasculitis in disease remission (Experimental): * Participants will undergo a forearm blood flow study where forearm vasodilatation will be assessed in response to acetylcholine (7.5, 15 and 30ug/min) and sodium nitroprusside (1, 2 and 4ug/min).
  * Participants will also receive bradykinin (100, 300 and 1000pmol/min) in order to assess tPA release to measure fibrinolytic capacity.
  * Participants will also have 24-hour blood pressure measured, as well as measurements of arterial stiffness, choroidal volume and balance of peripheral inflammatory and anti-inflammatory cells.
  * After these baseline measurements have been obtained, the subject will receive 6 week of Bosentan. The participant will undergo the same investigations to compare if measurements differ after treatment.
  Interventions: Drug: Bosentan and dapagliflozin
- 30 age-, sex- and cardiovascular disease risk-matched control participants (No Intervention): * Participants will undergo a forearm blood flow study where forearm vasodilatation will be assessed in response to acetylcholine (7.5, 15 and 30ug/min) and sodium nitroprusside (1, 2 and 4ug/min).
  * Participants will also receive bradykinin (100, 300 and 1000pmol/min) in order to assess tPA release to measure fibrinolytic capacity.
  * Participants will also have 24-hour blood pressure measured, as well as measurements of arterial stiffness, choroidal volume and balance of peripheral inflammatory and anti-inflammatory cells.
  * These measurements will be compared to the large vessel vasculitis group to assess if there are differences in these measurements.

INTERVENTIONS:
Drug: Bosentan and dapagliflozin — Participants with LVV will receive Bosentan 62.5 mg twice daily and Dapagliflozin 10 mg once daily for 6 weeks, followed by Dapagliflozin 10 mg once daily for 4 weeks.
  Arms: 30 participants with large vessel vasculitis in disease remission

SUMMARY:
Large vessel vasculitis (LVV) is a disease that causes damage to blood vessels. This damage to blood vessels can increase the risk of patients with LVV developing cardiovascular disease, including heart attacks and strokes. A chemical produced in the body called endothelin may contribute to this increase in cardiovascular disease risk by causing the vessels to stiffen and blood pressure to increase.

It has previously been shown that by blocking the effects of endothelin, vessel stiffness and blood pressure improve. Bosentan is a tablet that blocks the effects of endothelin.

Dapagliflozin is a sodium-glucose co-transporter 2 inhibitor that has been shown to improve blood vessel function and stiffness in patients with diabetes.

The investigators plan to assess blood vessel function in those with LVV and participants without LVV. Participants with LVV will be given Bosentan and Dapagliflozin for 6 weeks, followed by Dapagliflozin for 4 weeks, to evaluate their impact on blood vessel function.

DETAILED DESCRIPTION:
Large vessel vasculitis (LVV) is an autoimmune disease characterised by inflammatory damage to the blood vessels. Although symptoms initially are non-specific, complications such as vessel stenosis can lead to heart failure and stroke. While current immunosuppressive treatments have improved short-term outcomes, they have not led to improvements in long-term outcomes. Patients with LVV remain at an increased risk of developing cardiovascular disease, the underlying mechanisms of which are not yet fully understood.

The inflammatory damage to blood vessels in LVV can result in endothelial dysfunction. Endothelin-1 (ET-1) is a potent vasoconstrictor produced by the endothelium. In endothelial dysfunction, excess ET-1 production causes raised blood pressure, increased arterial stiffness and reduced fibrinolytic capacity. Previous research has demonstrated that short-term blockade of endothelin receptors improves arterial stiffness and fibrinolytic capacity.

Inhibitors of the sodium-glucose co-transporter 2 (SGLT2i) target the renal proximal tubule to promote glycosuria. Recent large studies have demonstrated their impressive cardiovascular benefits across a range of conditions. Previous work has also demonstrated their ability to improve endothelial function and arterial stiffness in patients with diabetes.

Recently, the randomised, active-controlled Zenith-CKD trial demonstrated that the combination of zibotentan (an endothelin receptor antagonist) and the SGLT2 inhibitor dapagliflozin was effective in reducing albuminuria in patients with chronic kidney disease. Part of the rationale for combining these therapies was to offset the potential for fluid retention with zibotentan alone by harnessing the diuretic effect of dapagliflozin. The safety profile of an endothelin receptor antagonist and an SGLT2 inhibitor was excellent.

Bosentan is a dual endothelin receptor antagonist approved for the treatment of pulmonary arterial hypertension. Combining it with dapagliflozin will minimise the potential for fluid retention. Additionally, the potential for improved endothelial function and enhanced CVD protection with both of these agents used in combination is significant. To date, dual endothelin receptor antagonism and SGLT2 inhibition have not been trialled in patients with LVV.

The investigators will conduct a cross-sectional, case-control study comparing blood vessel function in patients with LVV with sex-, age-, and cardiovascular disease risk factor-matched control participants. This will be followed by an open-label trial in patients with LVV. Patients with LVV will be given 6 weeks of treatment with Bosentan and dapagliflozin, followed by 4 weeks of dapagliflozin to assess whether these drugs can improve blood vessel function and stiffness. Assessment of blood vessel function will be measured by venous occlusion plethysmography, a gold standard measure.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of large vessel vasculitis that has been in remission for ≥ 6 months.

Exclusion Criteria:

* Age <18 years
* Active LVV
* Any organ transplant recipients
* A requirement for any medications that are contra-indicated whilst taking Bosentan or dapagliflozin
* Congestive cardiac failure
* Patients not medically fit to attend study visits
* Patients without mental capacity or willingness to provide informed consent
* History of multiple and/or severe (clinical judgement as determined by the Investigator) allergic reactions to drugs, including the study drug, or food
* Patients who are pregnant or breast feeding, or those who plan to become pregnant during the study
* Participation in another clinical trial for 28 days before or 90 days after the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 6 in forearm blood flow | Before and after 6 weeks of treatment
  Change from baseline to week 6 in acetylcholine-mediated forearm blood flow vasodilation

SECONDARY OUTCOMES:
Change from Baseline to week 6 in fibrinolytic capacity | Before and after 6 weeks of treatment
  Plasma concentration of tissue plasminogen activator in response to bradykinin will be assessed before and after 6 weeks of intervention
Change from Baseline to week 6 in 24h blood pressure | Before and after 6 weeks of treatment
  24-hour ambulatory systolic and diastolic blood pressure will be assessed at baseline and 6 weeks.
Change from baseline to week 6 in arterial stiffness | Before and after 6 weeks of treatment
  Arterial stiffness will be assessed using pulse wave velocity as measured using SphygmoCor technology. Percentage change in pulse wave velocity will be compared between baseline and 6 weeks
Change from baseline to week 6 assessment of eye microvasculature using retinal OCT | Before and after 6 weeks of treatment
  Choroidal volume will be assessed using optical coherence tomography which will be compared at baseline and 6 weeks
Change from baseline to week 6 peripheral blood cells (balance of inflammatory and anti-inflammatory cells) analysed using flow cytometry | Before and after 6 weeks of treatment
  Flow cytometry will be used to assess peripheral blood cells (balance of pro-inflammatory and anti-inflammatory cells) at baseline and 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom